CLINICAL TRIAL: NCT02435069
Title: A Within Subjects Comparison of Two Antegrade Flushing Regimens in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Kim Jarczyk, Retired. Non-associate Emeritus, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ksj-1
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Fecal Incontinence; Neurogenic Bowel
Keywords: cecostomy; appendicostomy
MeSH Terms: conditions — Fecal Incontinence; Neurogenic Bowel | interventions — Sodium Chloride; Glycerol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pre-operative Baseline Phase (No Intervention): Baseline data including frequency and severity of fecal soiling and frequency and severity of abdominal pain were collected for a minimum of 2 weeks prior to surgical construction of the ACE stoma. Baseline stool calprotectin and serum electrolytes were collected in the baseline phase prior to initiation of the preoperative bowel prep. Pre-operative data served as the control.
- Dose Response - NS and USP Glycerin - First Intervention (Experimental): Initial flush used NS or USP Glycerin randomized to treatment sequence. The starting volume and administration frequency for NS was 10mL/kg and glycerin 20 mL administered every other day. The NS dose was titrated in 10 mL increments to achieve continence so as not to exceed 500 mL daily for a child under five years of age and 1000 mL daily for a child over 5 years of age. USP Glycerin was titrated in 5 mL increments so as not to exceed 50 mL daily. For side effects greater than Wong Bailey Faces Pain Rating Scale (WBFPRS) level 4, NS was decreased by 2.5 mL/kg to the lowest dose of 5 mL/kg daily. USP Glycerin was decreased in 5 mL increments to the lowest dose of 5 mL daily. If the maximum dose did not result in continence, if the dose necessary to minimize side effects resulted in fecal soiling, or if there were side effects greater than WBFPRS level 4 at the lowest dose of administration, the child was be trialed on the alternate therapy and then dropped from the study.
  Interventions: Drug: Dose Response - NS and USP Glycerin - First Intervention
- NS and USP Glycerin - Effectiveness - Second Intervention (Experimental): To prevent statistical bias from subject loss due to treatment failure, each child was randomized to a second treatment sequence once they achieved continence on optimal dosing with minimal side effects.This arm evaluated the long term effectiveness of NS and glycerin at optimal dose and administration frequency for 4 weeks and served as comparison between flush solutions. The study concluded with the child being placed back on 2 weeks of the initial flush in the randomized sequence.
  Interventions: Drug: Effectiveness - NS and USP Glycerin - Second Intervention

INTERVENTIONS:
Drug: Dose Response - NS and USP Glycerin - First Intervention — This trial used a repeated measures, single subjects alternating treatments A-B-C-B'-C'-B1' withdrawal design in which all subjects were tested under all conditions and each subject acted as his or her own control. The subjects were randomly assigned to either normal saline or USP glycerin to control for order effects. Baseline data A served as the control and was obtained pre-operatively. The B-C arm evaluated dose-response relationship and was used to identify the minimum dosing volume and frequency of ACE administration of NS and USP Glycerin necessary to promote fecal continence. When the optimal dose as identified, the child continued on that dose for 2 weeks to insure treatment stability and effectiveness.
  Other Names: 0.9% sodium chloride solution, Glycerol, Glycerin
  Arms: Dose Response - NS and USP Glycerin - First Intervention
Drug: Effectiveness - NS and USP Glycerin - Second Intervention — To prevent statistical bias from subject loss due to treatment failure, each child was randomized to a second treatment sequence once they have achieved continence with minimal side effects on optimal dosing The second phase B'-C'-B1' of the study compared the two regimens at optimal dose and administration frequency. This phase was used to confirm the effectiveness of NS and USP Glycerin at optimal dosing on continence and assess side effects.
  Other Names: 0.9% sodium chloride solution, Glycerol, Glycerin
  Arms: NS and USP Glycerin - Effectiveness - Second Intervention

SUMMARY:
There is a surgical procedure to help children with intractable fecal incontinence gain continence for stool through construction of a tube that connects the abdominal wall to the colon near or through the appendix. This tube allows easy administration of enema solution into the first part of the colon. Putting enema solution through that tube into the colon is called an antegrade continence enema (ACE) and has been shown to work well in helping some but not all children prevent stool accidents. The purpose of this study is to compare a large volume ACE flush using a salt water solution called normal saline with a small volume ACE flush using liquid glycerin. The aims of this study are to: 1) find the most effective dose and flush frequency of each solution needed to prevent stool accidents; 2) compare which solution given at the best dose has the least side effects and 3) to determine if administration of either of the ACE flushing solutions causes electrolyte abnormalities or affects colon health.

DETAILED DESCRIPTION:
Fecal incontinence past the time of toilet training is devastating to affected children. Antegrade continence enema (ACE) therapy administered through a catheterizable stoma surgically placed in the cecum has helped children with intractable fecal incontinence attain continence for stool. There are a number of retrospective studies demonstrating the variable effectiveness rates of ACE therapy. This variability may be due to what is used to flush. There are no prospective trials evaluating the effectiveness of different flushing regimens. The catheterizable stoma used for the antegrade administration of enema solution is frequently made by bringing the appendix out through the abdominal wall or by placing a skin-level device (button) in to the cecum. ACE therapy administration through the appendix or into the cecum has the potential to cause colonic dysfunction. The effects of ACE administration on colonic mucosal health has not been investigated. This pilot study will compare a high volume normal saline (NS) flush and a low volume United States Pharmacopeia (USP) glycerin flush. The primary aims of the study are to compare which solution, given at an optimal dose and frequency, is associated with fewer side effects, while promoting the higher degree of fecal continence, and to determine if antegrade enema solution administration through an appendicostomy/cecostomy causes electrolyte abnormalities or affects gut health.

ELIGIBILITY:
Inclusion Criteria:

* This study will involve twelve children ages 3 to 12 years recruited from subspecialty clinics at Nemours Children's Subspecialty Care and the Pediatric Spinal Defects Clinic in Jacksonville, Florida.
* Children will be selected by purposive sampling and will include those who are scheduled to have an ACE stoma and will require regular antegrade enema administration to maintain continence.

Exclusion Criteria:

* Excluded will be children with preexisting electrolyte imbalance, chronic high rectal tone, quadriplegia, renal or cardiac disease, or those who require prophylactic antibiotics, cannot communicate, or have significant cognitive delay that would interfere with their ability to fully participate in the study.
* Parents must have English language competency and be willing and able to participate in administration or oversight of the flushing regimen and data collection for a minimum of 20 consecutive weeks. -

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S Jarczyk, PhD, Principal Investigator — Nemours Children's Specialty Care
Locations (1):
- Nemours Children's Specialty Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksnes G, Diseth TH, Helseth A, Edwin B, Stange M, Aafos G, Emblem R. Appendicostomy for antegrade enema: effects on somatic and psychosocial functioning in children with myelomeningocele. Pediatrics. 2002 Mar;109(3):484-9. doi: 10.1542/peds.109.3.484. PMID 11875145
- [Background] Andersson RE, Olaison G, Tysk C, Ekbom A. Appendectomy is followed by increased risk of Crohn's disease. Gastroenterology. 2003 Jan;124(1):40-6. doi: 10.1053/gast.2003.50021. PMID 12512028
- [Background] Aspirot A, Fernandez S, Di Lorenzo C, Skaggs B, Mousa H. Antegrade enemas for defecation disorders: do they improve the colonic motility? J Pediatr Surg. 2009 Aug;44(8):1575-80. doi: 10.1016/j.jpedsurg.2008.11.061. PMID 19635308
- [Background] Bani-Hani AH, Cain MP, King S, Rink RC. Tap water irrigation and additives to optimize success with the Malone antegrade continence enema: the Indiana University algorithm. J Urol. 2008 Oct;180(4 Suppl):1757-60; discussion 1760. doi: 10.1016/j.juro.2008.04.074. Epub 2008 Aug 21. PMID 18721951
- [Background] Balter M. Taking stock of the human microbiome and disease. Science. 2012 Jun 8;336(6086):1246-7. doi: 10.1126/science.336.6086.1246. Epub 2012 Jun 6. No abstract available. PMID 22674333
- [Background] Bazar KA, Lee PY, Joon Yun A. An "eye" in the gut: the appendix as a sentinel sensory organ of the immune intelligence network. Med Hypotheses. 2004;63(4):752-8. doi: 10.1016/j.mehy.2004.04.008. PMID 15325028
- [Background] Becmeur F, Demarche M, Lacreuse I, Molinaro F, Kauffmann I, Moog R, Donnars F, Rebeuh J. Cecostomy button for antegrade enemas: survey of 29 patients. J Pediatr Surg. 2008 Oct;43(10):1853-7. doi: 10.1016/j.jpedsurg.2008.03.043. PMID 18926220
- [Background] Biglan A, Ary D, Wagenaar AC. The value of interrupted time-series experiments for community intervention research. Prev Sci. 2000 Mar;1(1):31-49. doi: 10.1023/a:1010024016308. PMID 11507793
- [Background] Chertow GM, Brady HR. Hyponatraemia from tap-water enema. Lancet. 1994 Sep 10;344(8924):748. doi: 10.1016/s0140-6736(94)92236-5. No abstract available. PMID 7915790
- [Background] Chow, S., & Liu, J. (2014). Design and analysis of clinical trials: Concepts and methodologies (3rd ed.). Hoboken, NJ: John Wiley & Sons.
- [Background] Chu DI, Balsara ZR, Routh JC, Ross SS, Wiener JS. Experience with glycerin for antegrade continence enema in patients with neurogenic bowel. J Urol. 2013 Feb;189(2):690-3. doi: 10.1016/j.juro.2012.08.209. Epub 2012 Oct 8. PMID 22986031
- [Background] Curry JI, Osborne A, Malone PS. The MACE procedure: experience in the United Kingdom. J Pediatr Surg. 1999 Feb;34(2):338-40. doi: 10.1016/s0022-3468(99)90204-x. PMID 10052818
- [Background] Dasso JF, Howell MD. Neonatal appendectomy impairs mucosal immunity in rabbits. Cell Immunol. 1997 Nov 25;182(1):29-37. doi: 10.1006/cimm.1997.1216. PMID 9427807
- [Background] Dey R, Ferguson C, Kenny SE, Shankar KR, Coldicutt P, Baillie CT, Lamont GL, Lloyd DA, Losty PD, Turnock RR. After the honeymoon--medium-term outcome of antegrade continence enema procedure. J Pediatr Surg. 2003 Jan;38(1):65-8; discussion 65-8. doi: 10.1053/jpsu.2003.50012. PMID 12592621
- [Background] Dolejs SC, Smith JK Jr, Sheplock J, Croffie JM, Rescorla FJ. Contemporary short- and long-term outcomes in patients with unremitting constipation and fecal incontinence treated with an antegrade continence enema. J Pediatr Surg. 2017 Jan;52(1):79-83. doi: 10.1016/j.jpedsurg.2016.10.022. Epub 2016 Oct 27. PMID 27817835
- [Background] Elder JH. Single subject experimentation for psychiatric nursing. Arch Psychiatr Nurs. 1997 Jun;11(3):133-8. doi: 10.1016/s0883-9417(97)80036-2. PMID 9193118
- [Background] Forchielli ML, Walker WA. The role of gut-associated lymphoid tissues and mucosal defence. Br J Nutr. 2005 Apr;93 Suppl 1:S41-8. doi: 10.1079/bjn20041356. PMID 15877894
- [Background] Gast, D.L. (2010). Single subjects research methodology in behavioral sciences. New York, NY: Routledge,Taylor & Francis Group
- [Background] Gebbers JO, Laissue JA. Bacterial translocation in the normal human appendix parallels the development of the local immune system. Ann N Y Acad Sci. 2004 Dec;1029:337-43. doi: 10.1196/annals.1309.015. PMID 15681775
- [Background] Gomez R, Mousa H, Liem O, Hayes J, Di Lorenzo C. How do antegrade enemas work? Colonic motility in response to administration of normal saline solution into the proximal colon. J Pediatr Gastroenterol Nutr. 2010 Dec;51(6):741-6. doi: 10.1097/MPG.0b013e3181e75d18. PMID 20890219
- [Background] Hartmann DP, Gottman JM, Jones RR, Gardner W, Kazdin AE, Vaught RS. Interrupted time-series analysis and its application to behavioral data. J Appl Behav Anal. 1980 Winter;13(4):543-59. doi: 10.1901/jaba.1980.13-543. PMID 16795632
- [Background] Helikson MA, Parham WA, Tobias JD. Hypocalcemia and hyperphosphatemia after phosphate enema use in a child. J Pediatr Surg. 1997 Aug;32(8):1244-6. doi: 10.1016/s0022-3468(97)90692-8. PMID 9269980
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Background] Ismail EA, Al-Mutairi G, Al-Anzy H. A fatal small dose of phosphate enema in a young child with no renal or gastrointestinal abnormality. J Pediatr Gastroenterol Nutr. 2000 Feb;30(2):220-1. doi: 10.1097/00005176-200002000-00025. No abstract available. PMID 10697146
- [Background] Janosky, J.E., Leininger, S.L., Hoerger, M.P., & Libkuman, T.M. (2009). Single subjects designs in biomedicine. New York, NY: Springer Science + Business Media.
- [Background] Janszky I, Mukamal KJ, Dalman C, Hammar N, Ahnve S. Childhood appendectomy, tonsillectomy, and risk for premature acute myocardial infarction--a nationwide population-based cohort study. Eur Heart J. 2011 Sep;32(18):2290-6. doi: 10.1093/eurheartj/ehr137. Epub 2011 Jun 1. PMID 21632600
- [Background] Jia W, Li H, Zhao L, Nicholson JK. Gut microbiota: a potential new territory for drug targeting. Nat Rev Drug Discov. 2008 Feb;7(2):123-9. doi: 10.1038/nrd2505. PMID 18239669
- [Background] Jones, B., & Kenward, M.G. (2003). Design and analysis of cross-over trials (2nd ed.). Boca Raton, FL: Chapman & Hall/CRC.
- [Background] Kaugars AS, Silverman A, Kinservik M, Heinze S, Reinemann L, Sander M, Schneider B, Sood M. Families' perspectives on the effect of constipation and fecal incontinence on quality of life. J Pediatr Gastroenterol Nutr. 2010 Dec;51(6):747-52. doi: 10.1097/MPG.0b013e3181de0651. PMID 20706148
- [Background] Kawanishi H. Immunocompetence of normal human appendiceal lymphoid cells: in vitro studies. Immunology. 1987 Jan;60(1):19-28. PMID 3493205
- [Background] Kazdin, A.E. (2011). Single-case research designs: Methods for clinical and applied settings (2nd ed.). New York, NY: Oxford University Press.
- [Background] King SK, Sutcliffe JR, Southwell BR, Chait PG, Hutson JM. The antegrade continence enema successfully treats idiopathic slow-transit constipation. J Pediatr Surg. 2005 Dec;40(12):1935-40. doi: 10.1016/j.jpedsurg.2005.08.011. PMID 16338323
- [Background] Knox CA, Burkhart PV. Issues related to children participating in clinical research. J Pediatr Nurs. 2007 Aug;22(4):310-8. doi: 10.1016/j.pedn.2007.02.004. PMID 17645958
- [Background] Large T, Szymanski KM, Whittam B, Misseri R, Chan KH, Kaefer M, Rink RC, Cain MP. Ambulatory patients with spina bifida are 50% more likely to be fecally continent than non-ambulatory patients, particularly after a MACE procedure. J Pediatr Urol. 2017 Feb;13(1):60.e1-60.e6. doi: 10.1016/j.jpurol.2016.06.019. Epub 2016 Aug 24. PMID 27614699
- [Background] Levitt MA, Soffer SZ, Pena A. Continent appendicostomy in the bowel management of fecally incontinent children. J Pediatr Surg. 1997 Nov;32(11):1630-3. doi: 10.1016/s0022-3468(97)90470-x. PMID 9396543
- [Background] Ma HH. An alternative method for quantitative synthesis of single-subject researches: percentage of data points exceeding the median. Behav Modif. 2006 Sep;30(5):598-617. doi: 10.1177/0145445504272974. PMID 16894232
- [Background] Marshall J, Hutson JM, Anticich N, Stanton MP. Antegrade continence enemas in the treatment of slow-transit constipation. J Pediatr Surg. 2001 Aug;36(8):1227-30. doi: 10.1053/jpsu.2001.25768. PMID 11479862
- [Background] Matsuno D, Yamazaki Y, Shiroyanagi Y, Ueda N, Suzuki M, Nishi M, Hagiwara A, Ichiroku T. The role of the retrograde colonic enema in children with spina bifida: is it inferior to the antegrade continence enema? Pediatr Surg Int. 2010 May;26(5):529-33. doi: 10.1007/s00383-010-2585-6. Epub 2010 Mar 3. PMID 20198477
- [Background] Nanigian DK, Nguyen T, Tanaka ST, Cambio A, DiGrande A, Kurzrock EA. Development and validation of the fecal incontinence and constipation quality of life measure in children with spina bifida. J Urol. 2008 Oct;180(4 Suppl):1770-3; discussion 1773. doi: 10.1016/j.juro.2008.03.103. Epub 2008 Aug 21. PMID 18721959
- [Background] Nicholson JK, Holmes E, Kinross J, Burcelin R, Gibson G, Jia W, Pettersson S. Host-gut microbiota metabolic interactions. Science. 2012 Jun 8;336(6086):1262-7. doi: 10.1126/science.1223813. Epub 2012 Jun 6. PMID 22674330
- [Background] National Institutes of Health. (1998). Policy on inclusion of children as research subjects in clinical research. Bethesda, MD: National Institutes of Health.
- [Background] Noverr MC, Huffnagle GB. Does the microbiota regulate immune responses outside the gut? Trends Microbiol. 2004 Dec;12(12):562-8. doi: 10.1016/j.tim.2004.10.008. PMID 15539116
- [Background] Ok JH, Kurzrock EA. Objective measurement of quality of life changes after ACE Malone using the FICQOL survey. J Pediatr Urol. 2011 Jun;7(3):389-93. doi: 10.1016/j.jpurol.2011.02.012. Epub 2011 Apr 27. PMID 21527223
- [Background] Peeraully MR, Lopes J, Wright A, Davies BW, Stewart RJ, Singh SS, More BB. Experience of the MACE procedure at a regional pediatric surgical unit: a 15-year retrospective review. Eur J Pediatr Surg. 2014 Feb;24(1):113-6. doi: 10.1055/s-0033-1357502. Epub 2014 Jan 17. PMID 24443094
- [Background] Penders J, Stobberingh EE, van den Brandt PA, Thijs C. The role of the intestinal microbiota in the development of atopic disorders. Allergy. 2007 Nov;62(11):1223-36. doi: 10.1111/j.1398-9995.2007.01462.x. Epub 2007 Aug 17. PMID 17711557
- [Background] Piantadosi, S. (2005). Clinical trials: A methodologic perspective (2nd ed.). Hoboken, NJ: John Wiley & Sons.
- [Background] Pieper P. Ethical perspectives of children's assent for research participation: deontology and on utilitarianism. Pediatr Nurs. 2008 Jul-Aug;34(4):319-23. PMID 18814566
- [Background] Polit, D.F. (2010). Statistical and data analysis for nursing research (2nd ed.). New York, NY: Pearson.
- [Background] Portney, L.G., & Watkins, M.P. (2009). Foundations of clinical research: Applications to practice (3rd ed.). Upper Saddle River, NJ: Pearson Prentice Hall.
- [Background] Randal Bollinger R, Barbas AS, Bush EL, Lin SS, Parker W. Biofilms in the large bowel suggest an apparent function of the human vermiform appendix. J Theor Biol. 2007 Dec 21;249(4):826-31. doi: 10.1016/j.jtbi.2007.08.032. Epub 2007 Sep 7. PMID 17936308
- [Background] Randall J, Coyne P, Jaffray B. Follow up of children undergoing antegrade continent enema: experience of over two hundred cases. J Pediatr Surg. 2014 Sep;49(9):1405-8. doi: 10.1016/j.jpedsurg.2014.02.090. PMID 25148747
- [Background] Rempher, K.J., & Silkman, C. (2007). How to appraise quantitative research articles. American Nurse Today, 2, 26-28.
- [Background] Schreiber CK, Stone AR. Fatal hypernatremia associated with the antegrade continence enema procedure. J Urol. 1999 Oct;162(4):1433; discussion 1433-4. doi: 10.1016/s0022-5347(05)68331-0. No abstract available. PMID 10492231
- [Background] Senn, S. (2002). Cross-over trials in clinical research (2nd ed.). West Sussex, England: John Wiley & Sons.
- [Background] Shuster, J.J. (2007). Design and analysis of experiments. In W.T. Ambrosius (Ed.). Topics in biostatistics (pp. 235-259). Totowa, NJ: Humana Press.
- [Background] Shuster JJ. Student t-tests for potentially abnormal data. Stat Med. 2009 Jul 20;28(16):2170-84. doi: 10.1002/sim.3581. PMID 19326398
- [Background] Siddiqui AA, Fishman SJ, Bauer SB, Nurko S. Long-term follow-up of patients after antegrade continence enema procedure. J Pediatr Gastroenterol Nutr. 2011 May;52(5):574-80. doi: 10.1097/MPG.0b013e3181ff6042. PMID 21502828
- [Background] Sinha CK, Grewal A, Ward HC. Antegrade continence enema (ACE): current practice. Pediatr Surg Int. 2008 Jun;24(6):685-8. doi: 10.1007/s00383-008-2130-z. Epub 2008 Apr 12. PMID 18408942
- [Background] Smith HF, Fisher RE, Everett ML, Thomas AD, Bollinger RR, Parker W. Comparative anatomy and phylogenetic distribution of the mammalian cecal appendix. J Evol Biol. 2009 Oct;22(10):1984-99. doi: 10.1111/j.1420-9101.2009.01809.x. Epub 2009 Aug 12. PMID 19678866
- [Background] Stenstrom P, Graneli C, Salo M, Hagelsteen K, Arnbjornsson E. Appendicostomy in preschool children with anorectal malformation: successful early bowel management with a high frequency of minor complications. Biomed Res Int. 2013;2013:297084. doi: 10.1155/2013/297084. Epub 2013 Sep 23. PMID 24175287
- [Background] Thomas JC, Dietrich MS, Trusler L, DeMarco RT, Pope JC 4th, Brock JW 3rd, Adams MC. Continent catheterizable channels and the timing of their complications. J Urol. 2006 Oct;176(4 Pt 2):1816-20; discussion 1820. doi: 10.1016/S0022-5347(06)00610-0. PMID 16945657
- [Background] Tiryaki S, Ergun O, Celik A, Ulman I, Avanoglu A. Success of Malone's antegrade continence enema (MACE) from the patients' perspective. Eur J Pediatr Surg. 2010 Nov;20(6):405-7. doi: 10.1055/s-0030-1265156. Epub 2010 Oct 15. PMID 20954103
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Vande Velde S, Van Biervliet S, Van Renterghem K, Van Laecke E, Hoebeke P, Van Winckel M. Achieving fecal continence in patients with spina bifida: a descriptive cohort study. J Urol. 2007 Dec;178(6):2640-4; discussion 2644. doi: 10.1016/j.juro.2007.07.060. Epub 2007 Oct 22. PMID 17945290
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] Yardley IE, Pauniaho SL, Baillie CT, Turnock RR, Coldicutt P, Lamont GL, Kenny SE. After the honeymoon comes divorce: long-term use of the antegrade continence enema procedure. J Pediatr Surg. 2009 Jun;44(6):1274-6; discussion 1276-7. doi: 10.1016/j.jpedsurg.2009.02.030. PMID 19524753
- [Background] Yerkes EB, Rink RC, King S, Cain MP, Kaefer M, Casale AJ. Tap water and the Malone antegrade continence enema: a safe combination? J Urol. 2001 Oct;166(4):1476-8. PMID 11547116
- [Background] Youssef NN, Barksdale Jr E, Griffiths JM, Flores AF, Di Lorenzo C. Management of intractable constipation with antegrade enemas in neurologically intact children. J Pediatr Gastroenterol Nutr. 2002 Apr;34(4):402-5. doi: 10.1097/00005176-200204000-00016. PMID 11930097
- [Result] Jarczyk, K.S. (2017). A within subjects comparison of two antegrade flushing regimens in children. University of Florida, Gainesville, FL. UFE0051658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from subspecialty clinics at Nemours Children's Clinic in Jacksonville, Florida between February 2016 and January of 2017
Pre-assignment Details: 9 assessed for eligibility, 4 excluded (3 did not meet inclusion criteria and 1 surgery date significantly delayed), 5 consented and randomized to treatment sequence in dosing phase (3 started on saline followed by USP Glycerin, 2 started on USP glycerin followed by saline).
Groups:
- No Intervention: Pre-operative Baseline Phase: Baseline data including frequency and severity of fecal soiling and frequency and severity of abdominal pain were collected for a minimum of 2 weeks prior to surgical construction of the ACE stoma. Baseline stool calprotectin and serum electrolytes were collected in the baseline phase prior to initiation of the preoperative bowel prep. Pre-operative data served as the control.
- Post-Operative Dose Response: NS Then USP Glycerin: Subjects randomized to treatment sequence. Arm evaluated dose-response relationship and was used to identify the minimum dosing volume and frequency of ACE administration for NS and USP glycerin necessary to meet outcome criteria. NS started at 10mL/kg administered every other day. Dose titrated to achieve continence so as not to exceed 500 mL NS daily for a child under five years of age, 1000 mL NS daily for a child over 5 years of age. Participant continued on effective dose for 2 weeks to insure treatment stability and effectiveness. If the maximum dose did not result in continence, if the dose necessary to minimize side effects resulted in episodes of fecal soiling, or if there were side effects greater than WBFPRS level 4 at the lowest dose of administration, the child was trialed on the alternate therapy and then dropped from the study.
- Post-Operative Dose Response: USP Glycerin Then NS: Subjects randomized to treatment sequence. Arm evaluated dose-response relationship and was used to identify the minimum dosing volume and frequency of ACE administration for USP glycerin and necessary to meet outcome criteria. Glycerin started at 20 mL administered every other day. Dose titrated to achieve continence so as not to exceed 50 mL daily. Participant continued on effective dose for 2 weeks to insure treatment stability and effectiveness. If the maximum dose did not result in continence, if the dose necessary to minimize side effects resulted in episodes of fecal soiling, or if there were side effects greater than WBFPRS level 4 at the lowest dose of administration, the child was trialed on the alternate therapy and then dropped from the study.
- Effectiveness Phase: NS Then USP Glycerin: To prevent statistical bias from subject loss due to treatment failure, each child who successfully completed the dosing phase was randomized to a second treatment sequence once they have achieved continence on optimal dosing with minimal side effects. This arm evaluated the long term effectiveness of NS at optimal dose and administration frequency for 4 weeks and served as comparison between flush solutions. The study concluded with the child being placed back on 2 weeks of the initial flush in the randomized sequence.
- Effectiveness Phase: USP Glycerin Then NS: To prevent statistical bias from subject loss due to treatment failure, each child who successfully completed the dosing phase was randomized to a second treatment sequence once they have achieved continence on optimal dosing with minimal side effects. This arm evaluated the long term effectiveness of USP glycerin at optimal dose and administration frequency for 4 weeks and served as comparison between flush solutions. The study concluded with the child being placed back on 2 weeks of the initial flush in the randomized sequence.
Period: Preoperative Baseline Phase
Arm/Group | No Intervention: Pre-operative Baseline Phase | Post-Operative Dose Response: NS Then USP Glycerin | Post-Operative Dose Response: USP Glycerin Then NS | Effectiveness Phase: NS Then USP Glycerin | Effectiveness Phase: USP Glycerin Then NS
Started | 5 | 0 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Response - First Intervention
Arm/Group | No Intervention: Pre-operative Baseline Phase | Post-Operative Dose Response: NS Then USP Glycerin | Post-Operative Dose Response: USP Glycerin Then NS | Effectiveness Phase: NS Then USP Glycerin | Effectiveness Phase: USP Glycerin Then NS
Started | 0 | 3 | 2 | 0 | 0
Completed | 0 | 2 | 1 | 0 | 0
Not Completed | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Period: Effectiveness - Second Intervention
Arm/Group | No Intervention: Pre-operative Baseline Phase | Post-Operative Dose Response: NS Then USP Glycerin | Post-Operative Dose Response: USP Glycerin Then NS | Effectiveness Phase: NS Then USP Glycerin | Effectiveness Phase: USP Glycerin Then NS
Started | 0 | 0 | 0 | 1 | 1
Completed | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | No Intervention: Pre-operative Baseline Phase
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 66.6 (29.3309)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 2
  Asian | 1
  Hispanic | 1
  African-American | 1
Region of Enrollment [Number; unit: participants]
  United States | 5
Cause of Neurogenic bowel [Number; unit: participants]
  myelomeningocele | 4
  Spinal Cord Trauma - MVA | 1
Patulent anus [Number; unit: participants] | 5
Ambulatory [Number; unit: participants]
  Ambulatory | 4
  Wheel Chair User | 1
Presence of Fecal Incontinence at Baseline [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Fecal Soiling - Number of Participants That Gained and Maintained Continence on Each Flushing Regimen
Description: Fecal soiling was defined as non-toilet elimination, which was tracked and documented by the parent/child as direct event recording and tallied as the number of pairs of underwear/protective undergarments soiled with stool per day. The purpose of this outcome measure was to document the number of individuals who gained continence on NS and USP glycerin. Descriptive statistics was limited to percentage of total participants who achieved continence on each flushing regimen. Data was calculated on the last data point in the final phase for both the NS and USP glycerin flush.
Time Frame: Data collection started following consent and procedural training and was collected daily from day 1 for the duration of the study, an average of 135 days.
Population: The data from a total of 5 participants were analyzed for each arm of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Continent on NS Antegrade Flush: Number of participants that gained and maintained continence on antegrade enema.
- Subjects Continent on USP Glycerin: Number of participants that gained and maintained continence on USP Glycerin antegrade enema.
Arm/Group | Subjects Continent on NS Antegrade Flush | Subjects Continent on USP Glycerin
Number analyzed (Participants) | 5 | 5
Participants | 1 | 4

2. Primary Outcome: Fecal Soiling - Quantitative Count Detailing the Number of Episodes of Fecal Incontinence Per Day on NS and USP Glycerin
Description: Fecal soiling was defined as non-toilet elimination, which was tracked and documented by the parent/child as direct event recording and tallied as the number of pairs of underwear/protective undergarments soiled with stool per day. Descriptive statistics included mean and standard deviation. Inferential statistical analysis was accomplished using a two-tailed, two-sample pooled variance t test with a significance level set at 0.05, calculated on the data from the last day of the completed NS and USP Glycerin phases of the study. Power analysis conducted using data from this study with α = 0.5, power of .80, correlation between two means of .598, and effect size of 1.554 estimated a sample size of 11 would be needed to minimize the risk of a Type II error to (20%).
Time Frame: Data collection began following consent and procedural training and was collected daily from day 1 for the duration of the study, an average of 135 days.
Population: The data from a total of 5 participants were analyzed for each arm of the study.
Measure: Mean (Standard Deviation); unit: underwear soiled/day
Units Other Than Participants: Fecal Soiling
Groups:
- Episodes of Fecal Incontinence on NS Antegrade Flush: Number of episodes of fecal soiling that occurred daily on NS flushing regimen
- Episodes of Fecal Incontinence on USP Glycerin Antegrade Flush: Number of episodes of fecal soiling that occurred daily on a USP Glycerin flushing regimen
Arm/Group | Episodes of Fecal Incontinence on NS Antegrade Flush | Episodes of Fecal Incontinence on USP Glycerin Antegrade Flush
Number analyzed (Participants) | 5 | 5
Number analyzed (Fecal Soiling) | 9 | 1
underwear soiled/day | 2 (1.87) | 0.2 (0.45)
Statistical Analysis 1: Comparison: Episodes of Fecal Incontinence on NS Antegrade Flush vs Episodes of Fecal Incontinence on USP Glycerin Antegrade Flush; Inferential statistical analysis was accomplished using a two-tailed, two-sample pooled variance t test with a significance level set at 0.05. and calculated on the data from the last day of the completed NS and USP Glycerin phases of the study. Power analysis conducted using data from this study with α = 0.5, power of .80, correlation between two means of .598, and effect size of 1.554 estimated a sample size of 11 would be needed to minimize the risk of a Type II error to (20%); Test type: Superiority; p = 0.069751, two-sample pooled variance t-test — significance level set at <0.05 a priori; Two-tailed

3. Secondary Outcome: NS and USP Glycerin Flush Solution Dosing Frequency Necessary to Achieve Continence
Description: Flush administration frequency necessary to achieve continence was recorded as a single measure per subject per flush solution obtained as the number of flushes in the last three days of each dosing phase and recorded as either daily (1), every other day (2), or every third day (3). The larger the value, the less frequent the flush, the better the clinical outcome. Dosing frequency was measured using direct observational recording completed by the parent or child. Descriptive analysis included mean, and standard deviation. Inferential statistical analysis was accomplished using a two-tailed, two-sample pooled variance t test with a significance level set at 0.05. Descriptive and inferential statistics were calculated on the data from the last day of the completed NS and USP Glycerin phases of the study.
Time Frame: Frequency of administration data was collected as the total number of flushes recieved over the last three days of each dosing phase for both NS and USP Glycerin and recorded as either daily (1), every other day (2), or every third day
Population: The data from a total of 5 participants were analyzed for each arm of the study.
Measure: Mean (Standard Deviation); unit: Flush administration/day
Groups:
- Dosing Frequency on NS: The minimum frequency with which the NS antegrade flush was administered during the dosing phase of the study necessary to gain and maintain continence. Data includes the maximum frequency of administration trialed in subjects who failed to gain continence on NS antegrade flush.
- Dosing Frequency on USP Glycerin: The minimum frequency with which the USP Glycerin antegrade flush was administered during the dosing phase of the study necessary to gain and maintain continence. Data includes the maximum frequency of administration trialed in subjects who failed to gain continence on USP GLycerin antegrade flush.
Arm/Group | Dosing Frequency on NS | Dosing Frequency on USP Glycerin
Number analyzed (Participants) | 5 | 5
Flush administration/day | 1 (0) | 1.6 (0.894)
Statistical Analysis 1: Comparison: Dosing Frequency on NS vs Dosing Frequency on USP Glycerin; Inferential statistical analysis was accomplished using a two-tailed, two-sample pooled variance t test with a significance level set at 0.05. and calculated on the data from the last day of the completed NS and USP Glycerin phases of the study; Test type: Superiority; p = 0.172, two-sample pooled variance t-test; two tailed

4. Secondary Outcome: Flush Volume
Description: Flush volume was measured in mL/flush using a graduated cylinder and recorded by the parent or child with each flush and later calculated in mL/kg. Data derived from the last flush of the completed dosing phase of both NS and USP Glycerin were used to calculate flush volume. Descriptive analysis included mean, median, range, and standard deviation. Reported data excludes subjects who failed to gain and maintain continence on either flushing regimen.
Time Frame: Data for analysis was collected from the last flush of the NS and USP Glycerin dosing phase of the study
Population: Subjects limited to those who gained continence (2 saline, 4 USP Glycerin). One subject gained and maintained continence on saline in both the dosing and maintenance phases of the study and one subject who gained continence during the dosing phase of the study but failed to maintain continence on saline during the maintenance phase of the study.
Measure: Mean (Standard Deviation); unit: mL/flush
Groups:
- Flush Volume of NS: Volume of flush solution administered during the last NS flush completed in the dosing phase of the study. Data from subjects who failed to gain and maintain continence during the dosing phase of the study on the maximum saline flush volume (500mL for subjects under 5 years of age and 1,000 mL for subjects over 5 years of age) are not included in the data. Data includes one subject who gained and maintained continence on saline in both the dosing and maintenance phases of the study, and one subject who gained continence during the dosing phase of the study but failed to maintain continence on saline during the maintenance phase of the study.
- Flush Volume of USP Glycerin: Volume of flush solution administered during the last USP Glycerin flush completed in the dosing phase of the study. Data from subjects who failed to gain and maintain continence on the maximum USP Glycerin flush volume (50mL) are not included in the data.
Arm/Group | Flush Volume of NS | Flush Volume of USP Glycerin
Number analyzed (Participants) | 2 | 4
mL/flush | 39.215 (12.424) | 1.475 (0.457)

5. Secondary Outcome: Number of Participants With Any Electrolyte Abnormality
Description: Evaluated impact of NS and USP Glycerin antegrade flush on serum electrolytes using a blood test called a Basic Metabolic Panel. Data analysis limited to percentage of subjects demonstrating any electrolyte abnormality on NS or USP glycerin.
Time Frame: Collection dates included a baseline sample (week 1) and at the completion of the dosing trail for both NS and USP glycerin for a total of 3 samples
Population: The data from a total of 5 participants were analyzed for each arm of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Elelctrolye Abnormalities on NS FLush: Number of participants who had abnormalities in Basic Metabolic Panel on NS antegrade flush
- Elelctrolye Abnormalities on USP Glycerin FLush: Number of participants who had abnormalities in Basic Metabolic Panel on USP Glycerin antegrade flush
Arm/Group | Elelctrolye Abnormalities on NS FLush | Elelctrolye Abnormalities on USP Glycerin FLush
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

6. Secondary Outcome: Change in Stool Calprotectin Levels Assessed Through Comparing Levels Obtained Following Completion of NS and USP Glycerin Dosing Phases With the Baseline Value For Each Subject
Description: Stool calprotectin was used to evaluate the impact of NS and USP Glycerin antegrade flush on colonic health. Calprotectin levels were obtained at baseline and following completion of the NS and USP Glycerin dosing phase of the study. Descriptive data analysis included mean and standard deviation for each flush regimen. Inferential statistical analysis was accomplished using a two-tailed, two-sample pooled variance t test with a significance level set at 0.05. Both descriptive and inferential data analysis was calculated on the difference in calprotectin levels between samples obtained at baseline and samples obtained following the completion of the NS and USP Glycerin flush (value at completion of dosing phase - baseline value). The assumption was the length of each dosing phase was sufficient to achieve a credible active washout period and therefore levels obtained at the end of a phase reflected flushing regimen effects colonic health regardless of flush order.
Time Frame: as for outcome 5
Population: The data from a total of 5 participants were analyzed for NS and 4 participants for USP Glycerin
Measure: Mean (Standard Deviation); unit: μg/g
Groups:
- Calprotectin Levels Following NS FLush: Calprotectin level from stool sample obtained at completion of the NS dosing phase compared to baseline.
- Calprotectin Levels Following USP Glycerin FLush: Calprotectin level from stool sample obtained at completion of the USP Glycerin dosing phase compared to baseline.
Arm/Group | Calprotectin Levels Following NS FLush | Calprotectin Levels Following USP Glycerin FLush
Number analyzed (Participants) | 5 | 4
μg/g | 133.7 (183.359) | 108 (113.874)
Statistical Analysis 1: Comparison: Calprotectin Levels Following NS FLush; Inferential statistical analysis was accomplished using a two-tailed, two-sample pooled variance t test with a significance level set at 0.05. and calculated on the data from the difference in calprotectin levels between samples obtained at baseline and samples obtained following the completion of the NS and USP Glycerin flush in the dosing phase of the study; Test type: Superiority; p = 0.8028, two-sample pooled variance t-test; two-sided

7. Secondary Outcome: Cramping With Flush
Description: Cramping with flush was measured using the Wong Baker Faces Pain Rating Scale (WBFPRS). The WBFPRS has undergone extensive testing and has well established psychometrics in the pediatric population. The scale ranges from 0 (very happy without pain) to 10 (the worse pain imaginable). Each pain level is associated with a facial expression. The child is asked to choose the face that best describes his/her level of discomfort (ordinal data). The parent was instructed to call if the child had flushing regimen-associated discomfort greater than a 4 on the WBFPRS. Documentation of pain severity was completed by the parent and child on a data-collection form at the time of occurrence. Descriptive statistics including mean and standard deviation. Inferential statistical analysis was accomplished using a two-tailed, two-sample pooled variance t test with a significance level set at 0.05. Descriptive and inferential statistics were calculated on the last data point in the dosing phase.
Time Frame: Data analysis was completed on data obtained during the last flush in both the NS and USP Glycerin dosing phase
Population: The data from a total of 5 participants were analyzed for each arm of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pain With NS Antegrade Flush Administration: Abdominal pain or cramping associated with NS flush as measured by the WBFPRS
- Pain With USP Glycerin Antegrade Flush Administration: Abdominal pain or cramping associated with USP Glycerin flush as measured by the WBFPRS
Arm/Group | Pain With NS Antegrade Flush Administration | Pain With USP Glycerin Antegrade Flush Administration
Number analyzed (Participants) | 5 | 5
units on a scale | 0 (0) | 0.4 (0.89)
Statistical Analysis 1: Comparison: Pain With NS Antegrade Flush Administration vs Pain With USP Glycerin Antegrade Flush Administration; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.346594, two-sample pooled variance t test; two tailed

8. Secondary Outcome: Number of Participants Experiencing Vagal Symptoms With Flush
Description: Vagal symptoms including nausea, vomiting, sweating, dizziness, and pallor were noted by the parent. The parent was instructed to call if the child had any vagal symptoms. Documentation of any vagal symptoms was completed by the parent and child on a data-collection form at the time of occurrence. Data was analyzed as a percentage of subjects experiencing vagal symptoms during flush with NS and USP glycerin.
Time Frame: Data collection started with the first flush administered following discharge from the hospital and was collected with every subsequent flush through completion of the study, an average of 115 days.
Population: The data from a total of 5 participants were analyzed for each arm of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Vagal Symptoms With NS FLush: Number of subjects experiencing vagal symptoms with antegrade administration of NS flush solution
- Vagal Symptoms With USP Glycerin Flush: Number of subjects experiencing vagal symptoms with antegrade administration of USP GLycerin flush solution
Arm/Group | Vagal Symptoms With NS FLush | Vagal Symptoms With USP Glycerin Flush
Number analyzed (Participants) | 5 | 5
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year 1 month
Groups:
- Vagal Symptoms With NS Flush: Number of subjects experiencing vasovagal symptoms (symptom complex including pallor, diaphoresis, dizziness, weakness, nausea, with or without syncope) with antegrade administration of NS flush solution
- Vagal Symptoms With USP Glycerin Flush: Number of subjects experiencing vasovagal symptoms (symptom complex including pallor, diaphoresis, dizziness, weakness, nausea, with or without syncope) with antegrade administration of USP Glycerin flush solution
Arm/Group | Vagal Symptoms With NS Flush | Vagal Symptoms With USP Glycerin Flush
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vagal Symptoms With NS Flush (N=5) | Vagal Symptoms With USP Glycerin Flush (N=5)
Vasovagal Response (Vascular disorders) | 0 (0) | 1 (1) — Symptom complex reported by parent including pallor, diaphoresis, dizziness, weakness, nausea, with or without syncope

LIMITATIONS AND CAVEATS:
Titration time to continence, procedural time, quality of life outcomes and microbiome sample analysis not reported due to limited number of subjects completing protocol. Study remained open without additional recruits until P.I. retirement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT02435069/Prot_SAP_001.pdf